CLINICAL TRIAL: NCT03573492
Title: Bedside Ultrasound in the Assessment of Deep Venous Thrombosis: Effectiveness of In-Person Versus Online Instruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mercy Health Ohio (Other)
Collaborators: Lake Erie College of Osteopathic Medicine (Other); Mercy Health (Other)
Responsible Party: Principal Investigator, Alex Daves, Principal Investigator, Mercy Health Ohio
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 17-017
Record Dates: First submitted 2018-05-22; First posted 2018-06-29 (Actual); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Educational Status

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In-Person Education by Ultrasonographer (Active Comparator): In-person education of the DVT scanning technique by an RDMS-certified ultrasonographer
  Interventions: Other: Education
- Online Education (EM Sono) (Active Comparator): Online lectures of DVT scanning technique by an Emergency Ultrasound fellowship director
  Interventions: Other: Education

INTERVENTIONS:
Other: Education — Type of teaching being assigned to student arms

SUMMARY:
This study will examine the effectiveness of pre-recorded instructional videos in the use of bedside ultrasonography to ascertain the presence of a lower extremity deep venous thrombosis (DVT) as compared to in-person lectures and hands-on training.

DETAILED DESCRIPTION:
This will be a single site prospective pilot study analyzing the agreement between the results of ED student bedside ultrasonography and radiology-performed ultrasonography. Medical students rotating at St Elizabeth Boardman Hospital in the emergency department from any U.S. medical school will be considered for enrollment. Once a rotation has been set up by the medical student and the medical student coordinator, they will be given information on the study being performed and asked if they will be interested. The medical student coordinator will provide them this information. They will be instructed to reply to the co-P.I. if they are interested in participating in the project and given the formal consent to review upon receipt of their affirmative response.

Potential study participants will be provided envelopes by the co-P.I. containing both the formal written consent to participate in the study as well as a short knowledge test of ultrasound technology and the DVT study itself. The student will be required to first sign the consent form, then take the examination and receive a failing score in order to participate in the study. This pre-test will be based heavily on the quizzes from the EMSono learning modules. Permission has been obtained by Dr. Robert Jones to use these questions as the basis for the pre-test examination. A passing score on the pre-test assessment will be considered to be 80% or higher. The assignment list will be computer-generated using the website www.randomizer.org. Students will be given their numeric randomization assignments based on the order in which they finish their exam, after those that pass are excluded. The exact methodology is described in https://www.randomizer.org/tutorial/lesson2.html. Utilizing this methodology, a randomly-generated value of 1 shall be online training, and 2 shall be in-person training.

The study itself shall consist of two arms separated by training. The patient inclusion criteria will not vary between the two arms, only the level of student training. Additional data will be obtained regarding study participants prior to the start of the study, including: training level, approximate number of lower extremity ultrasound studies performed by the participant in the past, overall ultrasound experience, and any formal sonographic education or credentialing.

In the first arm, participating students must have completed the "Practical Scanning" and "Lower Extremity DVT Ultrasound" modules contained within the EMSono online ultrasound instruction. In the second arm, participating student must have attended the in-person training that will be provided by an RDMS-certified ultrasonographer, Kathryn Gentile. The training will last approximately 4 hours in each training method and will include instruction on performing a B-mode compression test of the deep veins of the lower extremities to assess for presence or absence of DVT. There will be no significant difference in the approximate content covered in each training method. Each arm must pass a practical examination in which they must demonstrate basic proficiency in the use of the ultrasound device as well as the ability to obtain all views necessary for their examinations. Failure of the practical exam will result in exclusion from the remainder of the study. They will also be required to repeat the pre-test assessment which will be tracked for improvement from their first pre-test assessment. Both arms will have their pre-test assessment, training, and post-test practical examination monitored by the P.I., co-P.I., ultrasonographer, or another suitable proctor.

Emergency department patients whom the physician has a clinical suspicion for lower extremity DVT or PE and have intention of ordering formal radiology department performed ultrasound will be consented to also have a bedside ultrasound performed by study participant. This consent will be obtained by either the resident or attending physician providing the care of the patient; at which point, the physician will inform whatever student study participant is currently on shift in the department. If there are multiple student study participants present and on shift in the department, the physician must inform a student in an appropriate manner. If a student has already begun to see the patient that is to receive the DVT assessment, then they shall be the study participant selected. If no student has begun to see the patient, then the student with the fewest number of US DVT scans performed in the course of this study will be the study participant selected. If neither of these factors are definitive, then the ED physician shall decide the student to perform the examination via coin toss. If a physical coin is unavailable, then a smartphone coin toss app will be considered an acceptable alternative. The device utilized to obtain these exams shall be a Philips Lumify linear 12-4 MHz probe attached to a Samsung Galaxy View 19" tablet.

In each arm, each participant shall perform the examination according to the methods described by the teaching methods; including what veins are considered to be studied and what techniques to utilize in order to assess for the presence or absence of DVT. The study participant must perform the bedside ultrasound and record their results on a standardized document which will be placed in a locked box inside the department. The information recorded shall include: patient information, reason for exam, date and time of exam, extremity studied, technical limitations, number ultrasound for the study participant, and findings. Data on the form shall be standardized and in check-box form whenever possible to avoid ambiguity. This sheet will be completed and placed in the locked box prior to the patient receiving their formal radiology department performed examination, the timing of which will be verified by the resident or attending physician. At the completion of the study, all charts will be reviewed by the co-P.I. and the results provided on the sheet shall be compared to the results of the formal radiologic ultrasound and the data will be analyzed.

Of note, no treatment will be initiated based on the student ultrasound alone. If the suspicion remains very high and for some reason there is an urgent need to initiate treatment (e.g. admitted patient needing bridge orders), then the resident or attending must either perform an ultrasound exam themselves or must be able to interpret the images obtained by the formal study as the basis for treatment. If the patient is diagnosed with a PE prior to the formal study being completed, therapy will not be withheld until the formal US as it is clearly indicated in PE. Every attempt will be made to document this on the chart or paper form as applicable so that the chart can be reviewed more thoroughly for times of meds given/scans done and studies and be appropriately rejected if significant confounding exists, such as a positive DVT on student scan, initiation of anticoagulation for PE, then subsequent formal US negative for DVT. Further, although the diagnosis of DVT does exist across a spectrum, the presence of any thrombus on the formal radiological study is cause to initiate treatment, regardless of whether or not it is hemodynamically significant. As such, the positive presence of a thrombus will be treated as an affirmative result in both studies; and a negative result will be considered as a complete lack of any evidence for DVT.

Students in particular present a unique research opportunity, as there is little existing evidence on training truly naïve ultrasound users in the Emergency Department. Prior evidence has focused primarily on resident and attending training in the use of bedside ultrasound. Further, this study simultaneously represents a significant learning opportunity for students who choose to enroll, in addition to having routine access to the ultrasound equipment usually reserved for use by resident and attending physicians. The research goals of this study will be modeled after the studies that exist for physician training. Therefore, the investigators will conduct the study for a period of 12 months, aiming to obtain a minimum of 100 studies. There will be no upper bound on the number of examinations performed.

At the end of each rotation period, the studies will be collected from the locked box by the co-P.I. and the results of the formal radiological study will be compared to the results of the student-performed study. The paper studies from the locked box will then be transferred to a locked drawer within the locked EM resident's workroom. Only the P.I., co-P.I., applicable research assistant, and residency coordinator will have access to the locked drawer. These will then be transferred to a primary and backup encrypted flash drive in a spreadsheet file using the standardized results on the data collection sheet and the patient's visit number, so that the drive does not contain any identifiable PHI. The backup drive shall remain in the locked drawer. The research assistant shall be responsible for compiling this data on a semi-weekly basis as well as generation and maintenance of the data files on the encrypted flash drive. It is expected that this will data processing task will last for 5 hours every 2 weeks for the duration of the project at a cost of $20 per hour.

The data will be analyzed and relevant statistical analyses performed on the data to determine whether there is a statistically significant difference between the radiological study result and the student study result in each arm, as well as the comparison between the two arms. These analyses will be performed either by the P.I., co-P.I., or an appropriate research assistant utilizing SPSS or similar statistical analysis application to determine differences in sensitivity and specificity of exams grouped by training type. One training method will be considered as superior to the other only if the p value for this data is <0.05.

ELIGIBILITY:
Inclusion Criteria of students:

* Voluntary participation in the study
* Signed written informed consent
* Completion of all requirements for their respective arm of the study

Exclusion Criteria of students:

* Passing preliminary ultrasound knowledge test
* Prior education by EMSono or by an RDMS-certified ultrasonographer for the assessment of lower extremity DVT
* Rotation period less than 4 weeks

Inclusion Criteria of patients:

* Age 18 or greater
* Clinical suspicion of DVT or PE
* Hemodynamic stability
* Intact decision-making capacity
* Voluntary presentation to the ED
* Formal radiological lower extremity DVT study ordered by appropriate provider.

Exclusion Criteria of patients:

* Trauma or other anatomic abnormality
* Known DVT diagnosis within 48 hours
* History of chronic DVT
* Indwelling catheter or hemodialysis access in the extremity to be studied
* Refusal to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2018-12-05 (Actual); Study Completion 2018-12-05 (Actual)

PRIMARY OUTCOMES:
Superior education technique | 30 days
  Whether pre-recorded instruction is capable of providing sufficient education to ED medical students to obtain accurate diagnosis of DVT via ultrasonography or if in-person education should continue to be considered the standard of training. This will be assessed by calculating the sensitivity and specificity of each education technique compared to the "gold standard" of the formal DVT ultrasound by radiology.

CONTACTS AND LOCATIONS:
Locations (1):
- Mercy Health Youngstown, Youngstown, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided